CLINICAL TRIAL: NCT02699905
Title: Neutrophil FFA2/GPR43 Receptor Expression in Patients With the Diagnosis of Sepsis
Acronym: GPR43Sepsis
Status: Withdrawn | Type: Observational
Why Stopped: data was received from another source, therefore phlebotomy was not necessary
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Zyad J. Carr, M.D., Assistant Professor, Department of Anesthesiology & Perioperative Medicine, Milton S. Hershey Medical Center
Other Study IDs: STUDY00004607
Record Dates: First submitted 2016-03-01; First posted 2016-03-07 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Sepsis; Septic Shock; Multiple Organ Dysfunction; Intra-abdominal Sepsis
Keywords: Sepsis; Septic Shock; Multiple Organ Dysfunction; FFA2; GPR43
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 mL of whole blood drawn at four time intervals during the study. Blood is centrifuged and the Buffy coat separated and flash frozen in liquid nitrogen. Quantitative PCR analysis is then performed to assess the expression of FFA2/GPR43 at different time points in the patient's illness.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sepsis: Patients with the diagnosis of sepsis or septic shock
  Interventions: Other: phlebotomy
- Control: Healthy control with no evidence of active infection, or recent infection in the past 4 weeks.
  Interventions: Other: phlebotomy

INTERVENTIONS:
Other: phlebotomy — phlebotomy

SUMMARY:
This study seeks to elucidate the quantitative expression of G - protein receptor 43/free fatty acid (GPR43/FFA2) receptors in patients with the diagnosis of sepsis and specifically, its expression as it relates to the severity of sepsis. The investigators hypothesize that patients with more severe sepsis, as defined by a higher SOFA (Sequential Organ Failure Assessment Score), will have decreased expression of the GPR43/FFA2 as compared to patients with lower SOFA scores, consistent with a less exuberant immune response to infection.

Patients admitted to Penn State Hershey Medical Center with a diagnosis of sepsis of any cause will undergo blood testing of leukocytes to determine the expressed quantity of GP43 during standardized time points of their illness and recovery. No interventions will be made in the standard clinical management of the patient. Additionally, healthy volunteers will be recruited to exam baseline GPR43 receptor expression between sepsis and control groups.

DETAILED DESCRIPTION:
Despite advancements in recognition and treatment, sepsis continues to be a frequently fatal condition comprising 750,000 cases in the US with an estimated death rate of 28-38%. Bacterial sepsis complications are the result of a cascade of inflammatory mediators secondary to the immune system's recognition and response to invading bacteria, intracellular constituents and metabolites. Bacterial recognition results in the widespread activation of biological mediators essential to the immune response such as cytokines, chemokines, prostaglandins and reactive oxygen species. These compounds result in the activation and up-regulation of neutrophils, monocytes at the cellular level as well as the physiological changes of sepsis such as hyperpyrexia, vasodilation, and tachycardia. Despite this generally coordinated response, it is likely that marked complications are related to the sequela of the uncontrolled immune response leading to significant injury to the lungs (Acute Respiratory Distress Syndrome), and other organs (acute renal failure, shock liver). In addition, there is question that impairment of the gut mucosal barrier may result in translocation of bacteria and perpetuate the multiple organ failure.

G protein-coupled receptors (GPCRs) comprise one of the largest collections of transmembrane proteins in the mammalian genome. Recently, a subfamily of G protein coupled receptors have been identified that utilize short chain free fatty acids as ligands, FFA1 (GPR40), FFA2 (GPR43) and FFA3 (GPR41). Research has intimated that these receptors are involved in essential biological crosstalk between colonic bacteria, host and immune defenses. Although highly conserved in structure, members of this sub family demonstrate differences in fatty acid specificity, intracellular signaling mechanisms and tissue localization. Specifically, FFA2 (GPR43)4 expression has been shown to be expressed in higher magnitudes within immune cells, has been hypothesized to be involved in the modulation of pro- and anti-inflammatory mediators, such as prostaglandin E2 and is involved in neutrophil chemotaxis in mice. GPR43 is involved in the process of differentiation of progenitor immune cells into monocytes and macrophages, a key component of host defense. In addition, highly selective expression of GPR43 in polymorphonuclear cells point to strong role in chemotaxis and recruitment of immune cells to foci of bacterial infection. Short chain fatty acids also activate GPR43 receptors on intestinal epithelial cells with rapid production of secondary chemokine and cytokines after being challenged with inflammation and infection, and likely aid in the coordinated immune response. GP43 is likely an essential component of the phagocytic chemotaxis that maintains normal intestinal immune defense. In a model of acute colitis, GPR43 knockout mice demonstrated increased mortality. The authors concluded that GPR43 deficiency likely suppressed the role of immune cells within the gut immune milieu leading to death from sepsis related complications. Conversely, in a chronic colitis model, GPR43 deficient knockout mice demonstrated reduced colonic inflammation, without overwhelming infection, the authors concluded that GPR43 has an unfavorable role in the manifestation of chronic inflammatory conditions. These findings were confirmed with at least one later study. In humans, fetal membrane expression of GPR43 was higher in parturients in preterm labor with signs of infection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sepsis or septic shock
* Age greater than eighteen years old.
* Ability to give informed consent (as determined by the attending physician) or presence of designated healthcare proxy that can give informed consent.

Exclusion Criteria:

* Patients or designated healthcare proxy with the inability to give informed consent.
* Patients under the age of eighteen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with the diagnosis of sepsis or septic shock admitted to the intensive care unit at Penn State Hershey Medical Center, Hershey PA 17033.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Quantitative FFA2/GPR43 receptor expression as a function of SOFA score | Time of diagnosis, 24, 72, 168 hour intervals
  Quantitative expression of FFA2/GPR43 will be measured at specific time intervals and compared to SOFA score.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Covington DK, Briscoe CA, Brown AJ, Jayawickreme CK. The G-protein-coupled receptor 40 family (GPR40-GPR43) and its role in nutrient sensing. Biochem Soc Trans. 2006 Nov;34(Pt 5):770-3. doi: 10.1042/BST0340770. PMID 17052194
- [Background] Brown AJ, Goldsworthy SM, Barnes AA, Eilert MM, Tcheang L, Daniels D, Muir AI, Wigglesworth MJ, Kinghorn I, Fraser NJ, Pike NB, Strum JC, Steplewski KM, Murdock PR, Holder JC, Marshall FH, Szekeres PG, Wilson S, Ignar DM, Foord SM, Wise A, Dowell SJ. The Orphan G protein-coupled receptors GPR41 and GPR43 are activated by propionate and other short chain carboxylic acids. J Biol Chem. 2003 Mar 28;278(13):11312-9. doi: 10.1074/jbc.M211609200. Epub 2002 Dec 19. PMID 12496283
- [Background] Cox MA, Jackson J, Stanton M, Rojas-Triana A, Bober L, Laverty M, Yang X, Zhu F, Liu J, Wang S, Monsma F, Vassileva G, Maguire M, Gustafson E, Bayne M, Chou CC, Lundell D, Jenh CH. Short-chain fatty acids act as antiinflammatory mediators by regulating prostaglandin E(2) and cytokines. World J Gastroenterol. 2009 Nov 28;15(44):5549-57. doi: 10.3748/wjg.15.5549. PMID 19938193
- [Background] Vinolo MA, Ferguson GJ, Kulkarni S, Damoulakis G, Anderson K, Bohlooly-Y M, Stephens L, Hawkins PT, Curi R. SCFAs induce mouse neutrophil chemotaxis through the GPR43 receptor. PLoS One. 2011;6(6):e21205. doi: 10.1371/journal.pone.0021205. Epub 2011 Jun 15. PMID 21698257
- [Background] Sina C, Gavrilova O, Forster M, Till A, Derer S, Hildebrand F, Raabe B, Chalaris A, Scheller J, Rehmann A, Franke A, Ott S, Hasler R, Nikolaus S, Folsch UR, Rose-John S, Jiang HP, Li J, Schreiber S, Rosenstiel P. G protein-coupled receptor 43 is essential for neutrophil recruitment during intestinal inflammation. J Immunol. 2009 Dec 1;183(11):7514-22. doi: 10.4049/jimmunol.0900063. Epub 2009 Nov 16. PMID 19917676
- [Background] Masui R, Sasaki M, Funaki Y, Ogasawara N, Mizuno M, Iida A, Izawa S, Kondo Y, Ito Y, Tamura Y, Yanamoto K, Noda H, Tanabe A, Okaniwa N, Yamaguchi Y, Iwamoto T, Kasugai K. G protein-coupled receptor 43 moderates gut inflammation through cytokine regulation from mononuclear cells. Inflamm Bowel Dis. 2013 Dec;19(13):2848-56. doi: 10.1097/01.MIB.0000435444.14860.ea. PMID 24141712
- [Background] Kim MH, Kang SG, Park JH, Yanagisawa M, Kim CH. Short-chain fatty acids activate GPR41 and GPR43 on intestinal epithelial cells to promote inflammatory responses in mice. Gastroenterology. 2013 Aug;145(2):396-406.e1-10. doi: 10.1053/j.gastro.2013.04.056. Epub 2013 May 7. PMID 23665276
- [Background] Senga T, Iwamoto S, Yoshida T, Yokota T, Adachi K, Azuma E, Hamaguchi M, Iwamoto T. LSSIG is a novel murine leukocyte-specific GPCR that is induced by the activation of STAT3. Blood. 2003 Feb 1;101(3):1185-7. doi: 10.1182/blood-2002-06-1881. Epub 2002 Sep 19. PMID 12393494
- [Background] Le Poul E, Loison C, Struyf S, Springael JY, Lannoy V, Decobecq ME, Brezillon S, Dupriez V, Vassart G, Van Damme J, Parmentier M, Detheux M. Functional characterization of human receptors for short chain fatty acids and their role in polymorphonuclear cell activation. J Biol Chem. 2003 Jul 11;278(28):25481-9. doi: 10.1074/jbc.M301403200. Epub 2003 Apr 23. PMID 12711604
- [Background] Bindels LB, Dewulf EM, Delzenne NM. GPR43/FFA2: physiopathological relevance and therapeutic prospects. Trends Pharmacol Sci. 2013 Apr;34(4):226-32. doi: 10.1016/j.tips.2013.02.002. Epub 2013 Mar 13. PMID 23489932
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Result] Yao YM, Redl H, Bahrami S, Schlag G. The inflammatory basis of trauma/shock-associated multiple organ failure. Inflamm Res. 1998 May;47(5):201-10. doi: 10.1007/s000110050318. PMID 9657252
- [Result] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675